CLINICAL TRIAL: NCT05798936
Title: Comparative Study of Polidocanol and Absolute Alcohol for Percutaneous Ultrasound Guided Treatment of Benign Thyroid Cyst
Brief Title: Comparative Study of Polidocanol and Absolute Alcohol for Percutaneous us Guided Treatment of Benign Thyroid Cyst
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amna Ahmed Ali Ahmed, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: US in benign Thyroid cysts
Record Dates: First submitted 2023-02-14; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Benign Thyroid Nodule; Thyroid Lump; Thyroid Cyst
MeSH Terms: interventions — Polidocanol; Ethanol

STUDY DESIGN:
Intervention Model Description: Based on determining the main outcome variable, the estimated minimum required sample size is 30 patients (15 patient in each group).
  The sample was calculated using G*power software 3.1.9.2., based on the following assumptions: Main outcome variable is the difference between mean value of:
  Group (A): 15 patients will be treated by Ultrasound-Guided Percutaneous Polidocanol Injection Group (B): 15 patients will be treated by Ultrasound-Guided percutaneous ethanol injection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polidocanol group (Experimental): Polidocanol is injected in the thyroid cyst under ultrasound guidance.
  Interventions: Drug: Polidocanol
- Alcohol group (Experimental): Alcohol is injected in the thyroid cyst under ultrasound guidance.
  Interventions: Drug: Alcohol

INTERVENTIONS:
Drug: Polidocanol — Polidocanol is injected under complete aseptic conditions. Before the treatment the diameter and volume of each nodule is calculated. To prevent serious hemorrhage, vessels located along the approach route will be carefully evaluated by using Doppler US.
  Other Names: Polidocanol solution
  Arms: Polidocanol group
Drug: Alcohol — Alcohol is injected under complete aseptic conditions. Before the treatment the diameter and volume of each nodule is calculated. To prevent serious hemorrhage, vessels located along the approach route will be carefully evaluated by using Doppler US.
  Other Names: Alcohol Ethyl
  Arms: Alcohol group

SUMMARY:
This study aims to compare the efficacy and safety of ultrasound-guided percutaneous ethanol injection and percutaneous polidocanol injection for the treatment of benign cystic and predominantly cystic thyroid nodules.

DETAILED DESCRIPTION:
Thyroid nodules are characterized by excessive structural growth, functional transformation, and/or cystic degeneration of one or several areas within the gland. According to various studies, 15-30% of thyroid nodules are cystic or predominantly cystic. Around 5% of patients with thyroid nodules may experience compressive symptoms or cosmetic concerns, and treatment may be required in these cases.

Simple aspiration is generally the initial management for the purpose of diagnosis and cyst volume reduction. However, the recurrence rate has been reported to be high (40% to 59%), depending on the number of aspirations and extent of fluid evacuation. After simple fine-needle aspiration, most cystic lesions (around 80%) refill and enlarge over time.

Surgery is a long-established therapeutic option for benign thyroid nodules. However, the cost of thyroid surgery, risk of temporary or permanent complications, and impact on quality of life remain relevant concerns.

Ultrasound-guided percutaneous ethanol injection (PEI) The mechanism of ethanol sclerotherapy is that ethanol induces cellular dehydration and protein denaturation, which are followed by coagulation necrosis, reactive fibrosis, and small-vessel thrombosis.

As regard (PEI)Pain is the most common side effect, other mild side effects or complications occurred in small numbers of patients like: Facial flushing, Mild dizziness, Intracystic haemorrhage, drunken sense, Perithyroidal leakage. There are other side effects, including transient vocal cord palsy, respiratory distress requiring emergency surgical treatment, and venous thrombosis, in sporadic cases.

Percutaneous Polidocanol sclerotherapy (PPI) may be a potential alternative to ethanol for the treatment of benign cystic and predominantly cystic thyroid nodules.Polidocanol is a liquid detergent sclerosant developed in 1936 as a topical and local anaesthetic consisting of 95% hydroxy poly ethoxydodecane and 5% ethyl alcohol. It has been used as a treatment for hemorrhoidal disease, venous malformations, symptomatic hepatic cysts, renal cysts, gastric varices, and digital mucous cysts.

The mechanism of treating cyst is probably destroying endothelial cells of capsular wall which causes aseptic inflammation; thus endothelial tissue atrophies and cyst cavity adhere and occlude.

The side effects are mild including mild localized pain and mild or moderate fever after PPI. So, PPI could be a safe and effective alternative to treat benign cystic or predominant cystic thyroid nodules.

ELIGIBILITY:
Inclusion Criteria:

* Single cystic or predominantly cystic nodules.
* Pressure symptoms or cosmetic problems.
* No malignant or indeterminate cytologic results after ultrasound-guided fine-needle aspiration.
* Normal serum thyroid hormone levels

Exclusion Criteria:

* Association of a nodules showing malignant features on us examinations.
* Malignant or indeterminate cytologic results after ultrasound-guided fine-needle aspiration.
* Abnormal serum thyroid hormone levels

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Size of the thyroid cystic nodule after sclerosing agent injection (polidocanol versus alcohol) | 3 months
  Size of the thyroid cyst is measured by ultrasound after 3 months of sclerosing agent injection